CLINICAL TRIAL: NCT05442450
Title: Efficacy of Oral Semaglutide in Overweight or Obesity : Randomized Controlled Trial (OSO Study - Oral Semaglutide for Obesity)
Brief Title: Efficacy of Oral Semaglutide in Overweight or Obesity
Acronym: OSO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, Director Endoscopy (Center for Obesity and Metabolic Therapy), Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIG/IEC-BH@R 27 /05.2022-03
Record Dates: First submitted 2022-06-19; First posted 2022-07-05 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet+excercise+oral semaglutide (Experimental): Participants will receive individual counselling sessions for reduced-calorie diet and physical activity (with 150 minutes per week of physical activity, such as walking). Participants in this group will receive oral Semaglutide drug along with diet and exercise. Treatment will be initiated with the 3 mg once-daily dose. The dose will be increased to 7 mg and then maximum of 14mg per day in 2-4weeks interval based on your symptoms (nausea, vomiting, constipation etc)
  Interventions: Drug: oral semaglutide
- Diet+excercise (No Intervention): Participants in this group will receive individual counselling sessions for reduced-calorie diet and increased physical activity (with 150 minutes per week of physical activity, such as walking).

INTERVENTIONS:
Drug: oral semaglutide — Participants in Experimental group will receive oral Semaglutide along with diet and exercise. Treatment will be initiated with the 3 mg once-daily dose. The dose will be increased to 7 mg and then maximum of 14mg per day in 2-4weeks interval based on patient tolerance.
  Other Names: Rybelsus tablet
  Arms: Diet+excercise+oral semaglutide

SUMMARY:
All the eligible participants after screening will be randomized into two groups (Group 1 and 2) by block randomization (block size of 4 and 6) using computer generated random number. Randomization is performed by the individual not involved in the study.

Participants in both groups will receive individual counselling sessions to help them adhere to a reduced-calorie diet (500-kcal deficit per day relative to the energy expenditure estimated at the time) and increased physical activity (with 150 minutes per week of physical activity, such as walking). Both diet and activity will be recorded daily in a diary or by use of a smartphone application or other tools and were reviewed during counselling sessions. Participants in group 1 also receive oral Semaglutide along with diet and exercise. Treatment will be initiated with the 3 mg once-daily dose. The dose will be increased to 7 mg and then maximum of 14mg per day in 2-4weeks interval based on patient tolerance. Dose escalation schedule will be used to decrease the gastrointestinal side effects. Participants will be assessed for gastrointestinal complaints (nausea, vomiting) during escalation and follow-up. Once the desired dose is achieved, patient will remain at the maximum 14mg daily dose unless a reduction was warranted owing to problems with side effects. In such cases, investigators will reescalate the dose once symptoms are resolved or diminished.The absorption of oral Semaglutide is affected by food and fluid in the stomach, hence patients receiving oral Semaglutide will be instructed to take each tablet with up to 120 mL of water in the morning, in a fasting state, and a minimum of 30 min before the first meal of the day. Counselling will be done by a dietician or a similar qualified healthcare professional every 4th week via visits/phone contacts till the completion of the study. Participants have to physically visit the hospital at the end of 28 weeks for assessment.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive consenting patients of both genders with either a BMI of 30 or greater or a BMI of 27 or greater with one or more treated or untreated weight-related coexisting conditions (i.e., prediabetes, hypertension, dyslipidemia, obstructive sleep apnea, or cardiovascular disease).

Exclusion Criteria:

* • Diabetes mellitus

  * A glycated haemoglobin level of 48 mmol per mole (6.5%) or greater,
  * A history of chronic pancreatitis
  * Acute pancreatitis within 180 days before enrolment
  * Previous surgical obesity treatment
  * Use of antiobesity medication within 90 days before enrolment
  * Pregnancy and planning for pregnancy
  * Known malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving a reduction in body weight of 5% or more from baseline | seven months
  The proportion of patients achieving a reduction in body weight of 5% or more from baseline

SECONDARY OUTCOMES:
The percentage change in body weight from baseline to week 28 | Week 0 to week 28
  The percentage change in body weight will be compared between two groups.
Achievement of body weight reduction greater than or equal to 10% (Yes/No) | From baseline (week 0) to end of treatment (week 28) ]
  Count of participants
Change in waist circumference | baseline (week 0) to end of treatment (week 28)
  measured in cm
Change in body mass index (BMI) | baseline (week 0) to end of treatment (week 28)
  measured in kg/m^2
Change in systolic blood pressure | baseline (week 0) to end of treatment (week 28)
  measured in mmHg
Change in diastolic blood pressure | baseline (week 0) to end of treatment (week 28)
  measured in mmHg
Change in fasting serum insulin | baseline (week 0) to end of treatment (week 28)
  Ratio to baseline

CONTACTS AND LOCATIONS:
Overall Officials: chandana merugu, MD DM, Study Chair — Asian Institute of Gastroenterology Hospitals; pratik chhabra, MD, Study Director — Asian Institute of Gastroenterology Hospitals; Rakesh kalapala, MD DNB, Principal Investigator — Asian Institute of Gastroenterology Hospitals; Nitin Jagtap, MD DNB, Study Chair — Asian Institute of Gastroenterology Hospitals; Anand V Kulkarni, MD DM, Study Chair — Asian Institute of Gastroenterology Hospitals; Anudeep Katrevula, MD DM, Study Chair — Asian Institute of Gastroenterology Hospitals
Locations (1):
- Asian Institute of Gastroenterology hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
Individuals identity will not be disclosed

REFERENCES:
- [Derived] Katrevula A, Kalapala R, Agrawal S, Jagtap N, Chhabra P, Kulkarni AV, Merugu C, Katukuri GR, Duvvur NR. Oral semaglutide for weight loss and liver fibrosis in overweight and obesity: A randomized controlled trial. Indian J Gastroenterol. 2025 Oct 9. doi: 10.1007/s12664-025-01856-7. Online ahead of print. PMID 41066034